CLINICAL TRIAL: NCT06059924
Title: Does the Management of Anastomotic Leakage After Low Rectal Resection Affect the Long-term Oncological Outcome: A Retrospective Propensity Score Adjusted Cohort Study
Brief Title: Does the Management of Anastomotic Leakage After Low Rectal Resection Affect Survival
Acronym: ISRECLeak
Status: Completed | Type: Observational
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Ignazio Tarantino, Senior Physician, Cantonal Hospital of St. Gallen
Other Study IDs: ISREC leakage rectal resection
Record Dates: First submitted 2023-09-15; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Rectal Cancer; Anastomotic Leak
Keywords: Rectal cancer; Low rectal resection; Anastomotic leakage; ISREC-classification; Cancer-specific survival; Propensity score
MeSH Terms: conditions — Rectal Neoplasms; Anastomotic Leak

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- leak: Patients with diagnosed anastomotic leakage after low rectal resection for rectal cancer UICC stage I to III
  Interventions: Other: Anastomotic leakage
- noleak: Patients without anastomotic leakage after low rectal resection for rectal cancer UICC stage I to III

INTERVENTIONS:
Other: Anastomotic leakage — Anastomotic leakage was defined as a defect of the intestinal wall at the anastomotic site leading to a communication between the intra- and extraluminal compartments. It was diagnosed by clinical, laboratory, radiological (ultrasound, endosonography, computed tomography), endoscopic, and/or surgical findings.
  Groups: leak

SUMMARY:
The aim of this retrospective cohort-study is to assess the effects of AL and its severity divided according the ISREC-classification on the long-term oncological outcome.

DETAILED DESCRIPTION:
Rectal cancer is one of the most common malignancies in the world. Its costs and cancer-related mortality are increasing worldwide. The surgical treatment was revolutionized in recent years by the total mesorectal excision (TME) technique as well as the laparoscopic, robotic, and transanal approach. But anastomotic leakage (AL) remains one of the most feared complications after low rectal resection regarding postoperative morbidity and mortality as well as functional outcome. Several risk factors causing AL like low level of anastomosis, large tumor mass, male gender, smoking, perioperative bleeding, and preoperative radio-chemotherapy are known. Protective ileo- or colostomy formation and transanal tube placement may decrease the risk of AL and reduces the rate of reoperation due to AL. Diverting results of the association between AL and the long-term oncological outcome (local recurrence, systemic recurrence, survival) are described in the current literature.

The International Study Group of Rectal Cancer (ISREC) provides a classification of AL according to its clinical management:

* Grade A results in no change in patient's management
* Grade B requires active therapeutic intervention without re-laparotomy
* Grade C requires re-laparotomy

This classification allows a good stratification regarding postoperative morbidity and mortality. However, the association between the ISREC-classification of AL and the long-term oncological outcome is not yet clear.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving elective low anterior resection (LAR) between February 1991 and December 2020 at the Cantonal Hospital of St. Gallen

Exclusion Criteria:

* Other diagnosis than rectal cancer
* Discontinuity resection (no anastomosis)
* Emergency situation
* R1-resection
* Incomplete staging
* Metastatic cancer
* 30-day mortality
* Decline of a retrospective data analysis
* Secondary malignancy
* Age under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients operated at the Cantonal Hospital of St. Gallen
Sampling Method: Non-Probability Sample
Enrollment: 941 (Actual)
Dates: Start 1991-02-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Cancer-specific survival | 30 days postoperative to 5 years postoperative

SECONDARY OUTCOMES:
Overall survival | 30 days postoperative to 5 years postoperative
Disease-free survival | 30 days postoperative to 5 years postoperative
Recurrence-free survival | 30 days postoperative to 5 years postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Ignazio Tarantino, PD Dr. med., Principal Investigator — Klinik für Chirurgie, Cantonal Hospital of St. Gallen
Locations (1):
- Cantonal Hospital of St. Gallen, Sankt Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rahbari NN, Weitz J, Hohenberger W, Heald RJ, Moran B, Ulrich A, Holm T, Wong WD, Tiret E, Moriya Y, Laurberg S, den Dulk M, van de Velde C, Buchler MW. Definition and grading of anastomotic leakage following anterior resection of the rectum: a proposal by the International Study Group of Rectal Cancer. Surgery. 2010 Mar;147(3):339-51. doi: 10.1016/j.surg.2009.10.012. Epub 2009 Dec 11. PMID 20004450